CLINICAL TRIAL: NCT05791942
Title: UCLA Health Patient Health Maintenance Text Reminder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Richard K. Leuchter, MD, Clinical Instructor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MAPreminder1
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Health Maintenance; Diabetes; Cancer
Keywords: primary care; digital outreach
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel-arm randomized control trial
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Holdout Condition: No reminder (No Intervention): Eligible, randomized participants will receive no text message reminder.
- Control Reminder (Experimental): Eligible, randomized participants will receive a generic text message reminding them to close their outstanding health gap.
  Interventions: Behavioral: Reminder of preventive care measures
- Anecdote-based Reminder (Experimental): Eligible, randomized participants will receive a text message reminding them to close their outstanding health gap. This message will contain an anecdote of a patient whose cancer was caught early through similar, recommended preventive screenings.
  Interventions: Behavioral: Reminder of preventive care measures; Behavioral: Persuasion via anecdote
- Call-to-action Reminder (Experimental): Eligible, randomized participants will receive a text message reminding them to close their outstanding health gap. This message will prompt people to take care of the health gap right away before it slips their mind.
  Interventions: Behavioral: Reminder of preventive care measures; Behavioral: Behavioral: Action prompt

INTERVENTIONS:
Behavioral: Reminder of preventive care measures — The investigators will send randomized participants an SMS reminder encouraging them to click the provided link and close their outstanding, overdue preventive care measures.
  The provided link will take them to their MyChart login page; after logging in, they would see their personalized My Action Plan Letter detailing their personalized, overdue preventive care measures.
  Arms: Anecdote-based Reminder; Call-to-action Reminder; Control Reminder
Behavioral: Persuasion via anecdote — The message will contain an anecdote of a patient whose cancer was caught early through similar, recommended preventive screenings.
  Arms: Anecdote-based Reminder
Behavioral: Behavioral: Action prompt — The message will prompt people to take care of the health gap right away before it slips their mind.
  Arms: Call-to-action Reminder

SUMMARY:
This is a prospective randomized clinical trial evaluating how behaviorally-informed outreach text message reminders impact patient engagement with primary care. This prospective randomized control trial is being implemented in conjunction with UCLA Health's larger quality improvement initiative (the My Action Plan Quality Improvement Initiative) in order to improve primary care preventive measure completion rates.

DETAILED DESCRIPTION:
UCLA Health will launch an initiative called My Action Plan which is an outreach effort targeting the primary care patients at UCLA who have an outstanding, clinically indicated primary care preventative care gap (e.g., overdue colorectal cancer screening, outstanding diabetes tests) and aims at encouraging patients to complete their overdue health maintenance measures.

At the beginning of each month, identified UCLA Health primary care patients will be enrolled in a trial the investigators have pre-registered under the title "UCLA Health Patient Health Maintenance Outreach Text Message" and randomized to receive one of four text messages informing them that they have overdue health maintenance measures and urging them to take action to complete these measures. These text messages will contain a link to their MyChart patient portal account, specifically linking them to a My Action Plan electronic letter that will contain a personalized list of outstanding preventive care items and actionable steps to complete the items.

In March and April 2023, if participants do not open their My Action Plan electronic letter within 7 days after the initial outreach, they will be enrolled in the trial described in the current pre-registration. This trial will evaluate the effect of sending a text reminder about health gaps as well as compare the effectiveness of different outreach text reminders. Patients will be randomly assigned in a 1:1:1:1 ratio to either the holdout control condition (without a reminder) or one of the three reminder arms (receiving one of three text reminders 2 weeks after the initial outreach message). Additionally, within each text-reminder arm, patients will be randomized to one of three time slots for getting the reminder. The investigators will examine patients' interaction with these reminders and how that ultimately translates to them completing their indicated health maintenance measures.

The UCLA Department of Medicine (DOM) intends to roll out this QI initiative at the beginning of the 2023 calendar year and continue it for a span of at least 12 months. Each month, the initiative targets patients whose birthday falls into that month. This proposed trial will run for two months (March and April 2023).

Analysis Plan:

The investigators will utilize patient-level ordinary least squares (OLS) estimation, with statistical inferences based on model-robust standard errors. The primary model term will be indicator variables for arm assignment.

The analysis will adjust for sex, age, race/ethnicity, indicators for screenings/tests that patients are due for, and whether patients have upcoming primary care appointments. Missing covariate values will be handled by including 'unknown' indicators, along with mean imputation for quantitative covariates.

The investigators will use this dataset to address two separate research questions.

Research question 1: The investigators will compare the average of Arms 2-4 with Arm 1 to test the average effect of sending a text reminder. If the average effect is significant, the investigators will explore if Arms 2, 3, and 4 separately differ from Arm 1.

Research question 2: The investigators will compare Arm 3, Arm 4, with Arm 2 to test whether, compared to a simple (control) reminder, it is more effective to boost patients' intentions to close the health gap via an anecdote or to prompt patients to take actions quickly.

Exploratory analyses will investigate heterogeneous treatment effects by patients' baseline motivation (i.e., the extent to which patients seem to have some intentions to get the screenings/tests) in two ways. First, the investigators will use each patient's history of screenings/tests to construct a proxy for their baseline motivation to obtain the due screenings/tests. Specifically, the investigator will calculate, among all the screenings/tests that are included in the My Action Plan Initiative and that a patient was due for in the past few years (exact time window TBD based on data availability), what percentage was completed by the patient (as far as UCLA Health could tell). A higher percentage indicates a higher baseline motivation to get the screenings/tests patients are due for during the study period. Second, the investigators will obtain demographics and medical information that UCLA Health is willing to provide (e.g., gender, age, race/ethnicity, history of cancer and other pre-existing conditions, family cancer history, past adherence to screenings/tests that are included in the My Action Plan Initiative, past receipt of influenza vaccination, frequency of doctor visits; time window of these variables is TBD depending on data availability). With such information, the investigators will train an algorithm to predict patients' baseline motivation level using patients in the holdout condition (Arm 1) as the ground truth. Specifically, the investigators will take the aforementioned information about patients in Arm 1 as input, and use whether they complete any of the screenings/visits recommended in the My Action Plan letter within 6 months as the outcome measure. Then the investigators will apply the algorithm to all patients to predict their baseline motivation level. For both approaches, the proxy for baseline motivation (Approach 1) and the predicted baseline motivation level (Approach 2) will be used to analyze the heterogeneous treatment effects of (1) Arms 3 and 4 (vs. Arm 2) and (2) the combination of Arms 2 and 4 vs. Arm 1.

Additionally the investigators will investigate proxies for whether patients face structural barriers to get screenings/tests as moderators, including socioeconomic factors at the zipcode level, insurance type, proxies for accessibility to healthcare resources such as distance from UCLA Health clinics.

The investigators will also explore how the effect of text reminders varies across the three times of the day when the reminders will be sent.

ELIGIBILITY:
Inclusion Criteria:

1. Empaneled to UCLA Health DOM Primary Care
2. Has at least one overdue health maintenance measure that the My Action Plan initiative focuses on
3. Has an active MyChart status
4. Can accept SMS messages from UCLA Health
5. Has not opened the My Action Plan electronic letter within 7 days of initial outreach
6. Has a March or April Birthday

Exclusion Criteria:

1. Under the age of 18
2. Deceased patients
3. Hospice patients
4. Has opted out electronic communication (bulk messages, email, and/or text)
5. For the final analysis, the investigators will further exclude patients who have scheduled appointments for all screenings/tests or completed all screenings/tests prior to the date when they are supposed to receive the reminder from this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10583 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
MyChart letter opened | 1 week after getting the reminder
  Percentage of participants across the different arms who open their personalized My Action Plan letter on MyChart

SECONDARY OUTCOMES:
Opening link within SMS Text message | 1 week after getting the reminder
  Percentage of participants across the different reminder arms who click on the link in the reminder message
Direct scheduling appointment rate | Time Frame: 2 weeks after getting the reminder
  Rate of which eligible participants directly schedule an appointment for diabetic retinal exams, diabetes education, or breast cancer screening in order to complete these overdue screening/test(s). These screenings/tests have dedicated appointment resources that people can directly schedule for.
Rate of taking action for one overdue screening/test | Time Frame: 2 weeks after getting the reminder
  Rate of which participants schedule an appointment to complete their overdue screening/test or start the online tool for colorectal screening
Completion rate of one screening/test | Time Frame: 6 months after getting the initial outreach text message
  Rate of completion of at least one screening/test within the observation window.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health Department of Medicine, Quality Office, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make any individual participant data available.